CLINICAL TRIAL: NCT03522779
Title: Antioxidant Responses to Exercise and Cherry Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, Jamie Cooper, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003902
Record Dates: First submitted 2017-01-19; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High-fat meal + placebo (Placebo Comparator): Participants will complete a high-fat meal challenge with a placebo beverage.The placebo will be designed to match the tart cherry juice for volume and macronutrient content, but without the phytonutrient content of the tart cherries.The high-fat breakfast meal will consist of 2 Sausage Biscuits (McDonalds Corporation). Blood draws will then be obtained at 1, 2 and 3 hours postprandially for antioxidant and oxidative stress measurements.
  Interventions: Other: High-fat meal
- High-fat meal + tart cherry (Experimental): Participants will complete a high-fat meal challenge with a tart cherry juice concentrate. 60 mL of montmorency tart cherry concentrate will be diluted with 100 mL of water.The high-fat breakfast meal will consist of 2 Sausage Biscuits (McDonalds Corporation). Blood draws will then be obtained at 1, 2 and 3 hours postprandially for antioxidant and oxidative stress measurements.
  Interventions: Dietary Supplement: Tart cherry Juice; Other: High-fat meal
- Exercise + high-fat meal + placebo (Placebo Comparator): Participants will perform an acute bout of submaximal aerobic exercise 15 hours prior to the high-fat meal test. The exercise will consist of 30 minutes of treadmill running at 70% of each participants' calculated heart rate reserve. The following morning participants will complete a high-fat meal challenge with a placebo beverage.The placebo will be designed to match the tart cherry juice for volume and macronutrient content, but without the phytonutrient content of the tart cherries.The high-fat breakfast meal will consist of 2 Sausage Biscuits (McDonalds Corporation). Blood draws will then be obtained at 1, 2 and 3 hours postprandially for antioxidant and oxidative stress measurements.
  Interventions: Other: High-fat meal; Other: Exercise
- Exercise + high-fat meal + tart cherry (Experimental): Participants will perform an acute bout of submaximal aerobic exercise 15 hours prior to the high-fat meal test. The exercise will consist of 30 minutes of treadmill running at 70% of each participants' calculated heart rate reserve.The following morning participants will complete a high-fat meal challenge with a tart cherry juice concentrate. 60 mL of montmorency tart cherry concentrate will be diluted with 100 mL of water.The high-fat breakfast meal will consist of 2 Sausage Biscuits (McDonalds Corporation). Blood draws will then be obtained at 1, 2 and 3 hours postprandially for antioxidant and oxidative stress measurements.
  Interventions: Dietary Supplement: Tart cherry Juice; Other: High-fat meal; Other: Exercise

INTERVENTIONS:
Dietary Supplement: Tart cherry Juice — Tart cherry juice will be used to compare antioxidant and oxidative stress levels in human plasma following a high fat meal.
  Arms: Exercise + high-fat meal + tart cherry; High-fat meal + tart cherry
Other: High-fat meal — A high fat meal will be given to elicit postprandial oxidative stress.
Other: Exercise — The exercise will consist of 30 minutes of treadmill running at 70% of each participants' calculated heart rate reserve.
  Arms: Exercise + high-fat meal + placebo; Exercise + high-fat meal + tart cherry

SUMMARY:
To date, there are no published studies on the effects of tart cherry consumption on postprandial antioxidant and oxidative stress levels following a high-fat meal. Further, no one has looked at the effects of prior exercise on a high-fat meal that includes high phytonutrients like tart cherries. Therefore, the purpose of this study is to examine the effects of tart cherry consumption on antioxidant and oxidative stress levels in human plasma after consumption of a high-fat meal, as well as the postprandial impact of prior exercise in combination with tart cherry consumption on a high-fat meal.

DETAILED DESCRIPTION:
Study Design: This will be a single blinded, randomized, cross-over design in healthy humans. There will be four study visits for the four different treatments: 1) a high-fat meal alone, 2) a high-fat meal with tart cherry consumption, 3) prior exercise to a high-fat meal alone, and 4) prior exercise to a high-fat meal with tart cherry consumption. All participants will complete all 4 treatments in a random order. There will be a 7-day washout period between each visit.

Subjects: We will recruit 25 apparently healthy, physically active (structured exercise > 3h/week) adult men, ages 18-30 years. All subjects will be normal weight based on body mass index (BMI = 18-24.9kg/m2) or body composition (14-24% body fat). The IRB proposal has been submitted and will be reviewed this month. The entire study will take place at the CTRU and sample analysis will take place in the Dept. of Food Science and Technology.

Protocol: For 24h prior to testing, participants will be provided with all food and beverages. This will allow us to control their antioxidant intake prior to testing. The lead-in diet will be representative of a standard American diet and be low in total antioxidants. Estimated total daily energy needs will be based on each participants predicted resting metabolic rate and multiplied by a moderate physical activity value (1.65). Participants will consume all foods that are provided and no additional foods or beverages, may be consumed. Participants will arrive at the CTRU at 0700 hours in the fasted state (no food or drink for 8-12h) and will have abstained from exercise for 48h, unless participating in one of the 2 exercise treatment visits. Baseline measurements of height, weight, blood pressure, and body fat percentage will be taken. An intravenous catheter will be placed in the antecubital vein and a baseline sample will be taken.

Participants will then complete a high-fat meal challenge, either with or without tart cherries depending on their treatment visit. The meals will have tart cherry juice or a placebo consumed with a high-fat meal. The placebo will be designed to match the tart cherry juice for volume and macronutrient content, but without the phytonutrient content of the tart cherries. The high-fat breakfast meal will be a Sausage Biscuit and Hash Browns (McDonalds Corporation). Blood draws will then be obtained at 1, 2 and 3 hours postprandially for antioxidant and oxidative stress measurements.

Acute Exercise Protocol: Two of the four treatments will include an acute bout of submaximal aerobic exercise performed 15 hours (1600 hours; 4:00p.m.) prior to the high-fat meal test. The exercise will consist of 30 minutes of treadmill running at 70% of each participants' calculated heart rate reserve (HRR). This will be a supervised session where participants will wear a heart rate monitor. Participants will also be asked to give their ratings of perceived exertion every 10 minutes during the exercise bout. Participants will be instructed to consume the dinner meal provided to them after this exercise session is complete, which will also be 8-12h prior to the high-fat meal test.

Sample Analysis: Plasma will be tested for total anthocyanins content by HPLC-UV/VIS as well as HPLC-ESI-MS. Antioxidant capacity, oxidative stress measurements will be performed by H-ORACFL and FRAP assays.

ELIGIBILITY:
Inclusion Criteria:

* Males, 18-30 years old, with normal body weight based on body mass index (BMI=18-24.9kg/m2) or are of normal weight based on body composition analysis using the DXA (14-24% body fat). Must also participate in 3 or more hours per week of exercise with 1.5 or more of those hours being aerobic exercise.

Exclusion Criteria:

* Anyone with a chronic disease, medication use, digestive disorders, any supplement use, and anyone who will not consume tart cherry product. Anyone who is on a weight loss program, or planning to alter their current exercise program before the study would finish. Anyone who has lost or gained more than 5% of their body weight in the past 3 months. Anyone who has allergies to food, is vegan or vegetarian, or is on a medically prescribed diet.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Antioxidant levels | Change from baseline to 3 hours postprandially
  Plasma will be tested for total anthocyanins content by HPLC-UV/VIS as well as HPLC-ESI-MS. Antioxidant capacity measurements will be performed by FRAP assays.
Change in oxidative stress levels | Change from baseline to 3 hours postprandially
  Oxidative stress measurements will be performed by H-ORACFL assays.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Cooper, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia - Department of Foods and Nutrition, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.